CLINICAL TRIAL: NCT05575258
Title: The Effects of Agro-ecological Farming Systems on Human Health -- A Randomized Controlled Trial of Agro-ecologically vs Conventionally Produced Foods on Human Health Biomarkers
Brief Title: The Effects of Agro-ecological Farming Systems on Human Health
Acronym: AGROHEALTH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Collaborators: GreenAcres Foundation (Unknown)
Responsible Party: Principal Investigator, Stephanvanvliet, Principal Investigator, Utah State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 12519
Record Dates: First submitted 2022-05-31; First posted 2022-10-12 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Inflammatory Response
Keywords: Human Nutrition; Agro-ecology; Metabolomics; Human Health; Gut Microbiome; Agriculture

STUDY DESIGN:
Intervention Model Description: This work will utilize a randomized cross-over design to compare an agroecological vs conventional sourced diet, and determine their effects on inflammation and cardio metabolic health signatures in middle-aged adults (35-60 y old). Diets will be isocaloric and matched for macronutrient content, and consumed for 44 days each with a 14-day washout (habitual diet) period in between. Blood, urine, and stool samples will be obtained at baseline and after the dietary interventions, in addition to data about physical activity and questionnaires regarding quality of life.
  Participants will be asked to complete four testing visits throughout their participation in the study (pre and post visits for each of the diets, which are 44 days each). Participants will be blinded to the diet they are consuming.
Who Masked: Participant
Masking Description: Participants will be masked to the type of diet (Agroecological or Conventional) they are consuming.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1: Agro (Green) - Conventional (Yellow) (Active Comparator): First, the agro-ecological sourced diet will be consumed.
  Secondly, the conventional sourced diet will be consumed.
  Interventions: Other: 44-Day Diet Conventionally Sourced - YELLOW Diet; Other: 44-Day Diet Agro-Ecologically Sourced - GREEN Diet
- Sequence 2: Conventional (Yellow) - Agro (Green) (Active Comparator): First, the conventional sourced diet will be consumed.
  Secondly, the agro-ecological sourced diet will be consumed.
  Interventions: Other: 44-Day Diet Conventionally Sourced - YELLOW Diet; Other: 44-Day Diet Agro-Ecologically Sourced - GREEN Diet

INTERVENTIONS:
Other: 44-Day Diet Conventionally Sourced - YELLOW Diet — Food for the conventional diet will be sourced from local grocery stores (non-organic produce) around Logan, UT, USA.
Other: 44-Day Diet Agro-Ecologically Sourced - GREEN Diet — Food for the agro-ecological diet will be sourced predominantly from the Greenacres farm (Cincinnati, OH, USA) and a limited number of other retailers that sell select foods from agro-ecological producers (Seal the Seasons, General Mills, Pecan Shop, Sol Simple).

SUMMARY:
As concerns regarding the effects of agriculture on human and environmental health mount, a growing number of farmers are seeking ways to improve health from the ground up. A promising way by which a growing number of farmers are seeking to improve environmental health is by using agro-ecological practices (i.e., farming more closely in harmony with natural systems), which include practices such as multi-cropping, ley rotations, and/or integrated crop-livestock systems. Despite potential ecological benefits, there is a lack of critical knowledge if consuming foods from agro-ecological systems impacts biomarkers of human health, including inflammatory and metabolomics profiles. The purpose of this project is to test the hypothesis that consuming foods produced using agro-ecological practices improves biomarkers of consumer health compared to consuming similar foods from conventional (monoculture) agriculture. All diets will be matched one-to-one in terms of macronutrients and food sources.

DETAILED DESCRIPTION:
This work will utilize a randomized cross-over design to compare an agroecological vs conventional sourced diet, and determine their effects on inflammation and cardio metabolic health signatures in middle-aged adults (35-60 y old). Diets will be isocaloric and matched for macronutrient content, and consumed for 44 days each with a 14-day washout (habitual diet) period in between. Blood, urine, and stool samples will be obtained before and after the dietary interventions, in addition to data about physical activity and questionnaires regarding quality of life.

STUDY OBJECTIVES

1. To determine the effects on plasma inflammatory markers (IL-6, TNF-α, C-reactive protein) in response to each intervention.
2. To determine effects on urinary and plasma metabolites (vitamin and mineral derivatives, polyphenols, amino acids, glucose metabolites etc.) to provide insight into metabolic health pathways in response to each intervention.
3. To determine effects on gut microbiota communities (alpha and beta diversity, and short-chain fatty acid producing bacteria) in response to each intervention.

INTERVENTION

After completing all baseline testing, participants will be randomized to one of the two starting diets (agroecological or conventional, for 44 days with a 14 day washout period until they start their second diet (agroecological or conventional depending on the starting diet). In accordance with established protocols, a research dietitian will provide weight-maintenance diets based on each individual's daily energy requirement (Harris-Benedict equation). All foods that participants consume during those 44 days will be provided by the Metabolic Kitchen at NDFS, and dietitian-led group classes and handouts with food preparation instructions will be provided to the participants to ensure compliance. The diets will be provided as 4-day rotating menus and participants will be asked to pick-up food twice weekly at the NDFS building. This will allow the research time to interact face-to-face with the participant, address any issues, and further ensure compliance. All subjects assigned to the same diet will receive identical meals and snacks, but portion sizes will be determined based on the previously mentioned daily energy requirement. Food for the agroecological diet will be sourced predominantly from the Greenacres farm (Cincinnati, OH) and/or other producers that use documented agro-ecological principles (e.g., Regenerative Organic Certified). Food for the conventional diet will be sourced from local grocery stores in Logan, UT (non-organic produce). All foods will be stored in food-grade fridges and freezers in the CHNS Metabolic Kitchen and food boxes will be prepared weekly by staff.

Examples of Meals

Breakfast Whole milk, eggs, oatmeal, and blueberries

Snack Rice cakes

Lunch Ground beef, tomato salad and cherries

Snack Apple with nut butter

Dinner Grilled chicken with rice and steamed broccoli

ELIGIBILITY:
Inclusion Criteria:

* Age ≥35 and ≤60 years
* BMI ≥25 and ≤35kg/m2
* Weight stable in last 3 months (loss or gain <4%)
* Hemoglobin A1C (HbA1C ≤6.4%)
* Fasting plasma glucose concentration <126mg/dl
* For the safety of the participant and proper consent of the procedures, subjects must be able to speak and understand English to participate in this study
* Stable medication/supplement use for 3 months prior to study

Exclusion Criteria:

* Use of medications that are known to affect the study outcome measures (e.g., NSAIDs, corticosteroids) or increase the risk of study procedures (e.g., anticoagulants) that cannot be temporarily discontinued for this study
* Strict dietary patterns (e.g., vegan, keto)
* Consuming >14 alcoholic drinks per week
* Use of cigarettes (or other tobacco products) in last 3 months
* Engaged in high level of competitive exercise (e.g., iron man, marathons, powerlifting)
* Diagnoses of active malignancy, congestive heart failure, diabetes mellitus or chronic obstructive pulmonary disease
* Any inflammatory diseases(e.g., autoimmune diseases, coeliac disease, glomerulonephritis, hepatitis, inflammatory. bowel disease, arthritis)
* Use of antibiotics in last 60 days
* Pregnant or planning to become pregnant in the next 5 months
* Lactating women
* Persons who are unable or unwilling to follow the study protocol or who, for any reason, the research team considers not an appropriate candidate for this study, including non-compliance with screening appointments or study visits
* Participants that are pregnant or planning on becoming pregnant in the next 5 months are excluded. The justification is the documented alterations in metabolism that occur during pregnancy, which would impact our metabolomics analysis in this study.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Inflammatory cytokine biomarker (IL-6 and TNF-alpha) concentrations in plasma samples | Day 44 (post)
  Inflammatory biomarker concentrations of IL-6 and TNF-alpha (pg/ml) will be measured using ELISA kits at the Center for Human Nutrition Studies at Utah State University. Blood samples will be obtained via phlebotomy at day 44 (post-diet) for each intervention, centrifuged immediately and stored at -80ºC until analyses are performed.
Inflammatory cytokine biomarker (C-reactive protein) concentrations in plasma samples | Day 44 (post)
  Inflammatory biomarker concentrations of C-reactive protein (CRP; ng/ml) will be measured using ELISA kits at the Center for Human Nutrition Studies at Utah State University. Blood samples will be obtained via phlebotomy on day 44 (post-diet) for each intervention, centrifuged immediately and stored at -80ºC until analyses are performed.
Relative abundance of metabolites in plasma samples using triple quad LC/MS-MS | Day 44 (post)
  Relative abundance (arbitrary units) of plasma metabolites after each diet will be measured using high-performance liquid chromatography tandem mass-spectrometry (LC/MS-MS). This analysis allows the simultaneous high-resolution measurement of a broad range of metabolites and will give insight into how food-derived metabolites from the two different diets impact metabolic pathways of human health. Blood samples will be obtained via phlebotomy on day 44 (post-diet) for each intervention, centrifuged immediately and stored at -80ºC until analyses are performed. Multivariate statistical analysis and Partial least squares Discriminant Analysis will be used to identify features change from pre to post on each diet.
Composition of gut microbiota bacteria using 16s rRNA sequencing | Day 44 (post)
  First of the day stool samples will be collected on day 44 (post-diet) for each intervention using DNA Genotek OMR-200 collection kits and stored at -80ºC until analyses are performed. DNA will be extracted from stool samples using a QIAamp Fast DNA Stool Mini Kit following manufacturer's instructions and analyzed for taxonomic assignment using 16s rRNA sequencing. Reported outcomes include individual bacteria and Shannon Index Values.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) scores | Day 44 (post)
  The PSQI will be used to determine sleep quality. Assessments will be performed on day 44 (post-diet) for each intervention. PSQI yields a total score ranging from 0 to 21 with a higher total score (referred to as global score) indicating worse sleep quality.
The Perceived Stress Scale (PSS) scores | Day 44 (post)
  PSS evaluates how unpredictable, uncontrollable, and overloaded participants judge their lives. Assessments will be performed on day 44 (post-diet) for each intervention. PSS scores can range from 0 to 40 with higher scores indicating higher perceived stress.
Profile of Mood States (POMS) scores | Day 44 (post)
  The Profile of Mood States (POMS) 30-item version will determine mood changes using the following domains: Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia and Confusion-Bewilderment. Assessments will be performed on day 44 (post-diet) for each intervention. This will give a value between -24 and 177, with lower scores indicative of people with more stable mood profiles.
Short Form Healthy Survey (SF-36) scores | Day 44 (post)
  The SF-36 will be used to assess quality of life using physical (functioning, role-physical, pain, general health) and mental domains (vitality, social functioning, role-emotional, and mental health). Assessments will be performed on day 44 (post-diet) for each intervention. The SF-36 scores on a range from 0-100 with higher scores indicating better physical and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan van Vliet, Principal Investigator — Utah State University
Locations (1):
- Center for Human Nutrition Studies, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Decoded metabolomics data will be posted in public repositories (Metabolomics Workbench)
  Decoded inflammatory biomarker, gut microbiome, and bloodwork data will be added as supplemental information to the publication.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: After analysis and publication are complete.

REFERENCES:
- [Background] Kronberg SL, Provenza FD, van Vliet S, Young SN. Review: Closing nutrient cycles for animal production - Current and future agroecological and socio-economic issues. Animal. 2021 Dec;15 Suppl 1:100285. doi: 10.1016/j.animal.2021.100285. Epub 2021 Jul 24. PMID 34312093
- [Background] Wezel, A.et al.Agroecological practices for sustainable agriculture. A review. Agronomy for Sustainable Development34, 1-20, doi:10.1007/s13593-013-0180-7 (2014).
- [Background] Albizua, A., Williams, A., Hedlund, K. & Pascual, U. Crop rotations including ley and manure can promote ecosystem services in conventional farming systems. Applied Soil Ecology95, 54-61, doi:https://doi.org/10.1016/j.apsoil.2015.06.003(2015).
- [Background] McDaniel MD, Tiemann LK, Grandy AS. Does agricultural crop diversity enhance soil microbial biomass and organic matter dynamics? A meta-analysis. Ecol Appl. 2014 Apr;24(3):560-70. doi: 10.1890/13-0616.1. PMID 24834741
- [Background] Lain KY, Catalano PM. Metabolic changes in pregnancy. Clin Obstet Gynecol. 2007 Dec;50(4):938-48. doi: 10.1097/GRF.0b013e31815a5494. PMID 17982337
- [Background] Galie S, Garcia-Gavilan J, Papandreou C, Camacho-Barcia L, Arcelin P, Palau-Galindo A, Rabassa A, Bullo M. Effects of Mediterranean Diet on plasma metabolites and their relationship with insulin resistance and gut microbiota composition in a crossover randomized clinical trial. Clin Nutr. 2021 Jun;40(6):3798-3806. doi: 10.1016/j.clnu.2021.04.028. Epub 2021 Apr 27. PMID 34130026
- [Background] Meslier V, Laiola M, Roager HM, De Filippis F, Roume H, Quinquis B, Giacco R, Mennella I, Ferracane R, Pons N, Pasolli E, Rivellese A, Dragsted LO, Vitaglione P, Ehrlich SD, Ercolini D. Mediterranean diet intervention in overweight and obese subjects lowers plasma cholesterol and causes changes in the gut microbiome and metabolome independently of energy intake. Gut. 2020 Jul;69(7):1258-1268. doi: 10.1136/gutjnl-2019-320438. Epub 2020 Feb 19. PMID 32075887
- See also: Google Scholar - Stephan van Vliet — https://scholar.google.com/citations?user=L5KcySQAAAAJ&hl=en
- See also: Center for Human Nutrition Studies - USU — https://caas.usu.edu/facilities/human-nutrition-studies

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT05575258/Prot_SAP_ICF_000.pdf